CLINICAL TRIAL: NCT05551689
Title: Evaluation of the Effectiveness of the FOCUS ADHD Mobile Health Platform in the Monitoring of Adults With Attention-Deficit/ Hyperactivity Disorder (ADHD)
Brief Title: FOCUS ADHD Mobile Health App for Adult ADHD Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2021-0084
Record Dates: First submitted 2022-09-16; First posted 2022-09-23 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: ADHD
Keywords: mhealth; app
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Alzheimer Disease | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Intervention Model Description: randomized clinical trial
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Participants are randomized by an independent assistant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ADHD monitoring as usual (Active Comparator): ADHD patient monitoring as usual based on psychostimulant prescription and follow up
  Interventions: Drug: Psychostimulant
- FOCUS ADHD (Experimental): ADHD patient monitoring as usual based on psychostimulant prescription and follow up plus the indication to use the FOCUS ADHD app as a treatment monitoring tool
  Interventions: Drug: Psychostimulant; Device: FOCUS ADHD App
- FOCUS ADHD and the elegibility for discount concession on treatment purchase (Experimental): ADHD patient monitoring as usual based on psychostimulant prescription and follow up plus the indication to use the FOCUS ADHD app as a treatment monitoring tool. In this arm patients are also eligible for a discount of at least 25% of the drug cost (after the first month of treatment) if they register and maintain at least 80% of their treatment adherence on the FOCUS ADHD app. The discount is granted after week 4 until the end of the follow up period.
  Interventions: Drug: Psychostimulant; Device: FOCUS ADHD App

INTERVENTIONS:
Drug: Psychostimulant — All enrolled patients should be receiving ADHD pharmacological treatment (psychostimulants)
  Other Names: Methilphenidate; Lisdexamfetamine
Device: FOCUS ADHD App — FOCUS ADHD is a mobile health application to support ADHD treatment adherence, monitoring and psychoeducation. The App was developed by the Attention Deficit Hyperactivity Disorder Program (ProDAH) of the Hospital de Clínicas de Porto Alegre (HCPA) and the Federal University of Rio Grande do Sul (UFRGS)
  Other Names: mhealth app
  Arms: FOCUS ADHD; FOCUS ADHD and the elegibility for discount concession on treatment purchase

SUMMARY:
The study is a randomized clinical trial to evaluate the efficacy on treatment adherence, performance and usability of the mobile health solution FOCUS ADHD, in combination with a discount application in the purchase of psychostimulant medication by adult patients with ADHD

DETAILED DESCRIPTION:
Current technological and digital advances enable the development and implementation of innovative and effective strategies in the diagnosis, treatment, and follow-up of patients with ADHD and other mental disorders. Such tools have the potential to significantly improve the services provided with a patient-centred approaches, expand and facilitate access to and support for treatment of adults with ADHD and other mental disorders. However, the levels of scientific evidence of such solutions are still limited and more studies are needed for their evaluation in different contexts and populations. The expectation is that such mHealth devices can help in the diagnosis, identification, and early detection of individuals at higher risk, allowing the development of individualized and more efficient approaches. At the same time, offering integrated, multidisciplinary, continuous, and accurate monitoring.

This project aims to evaluate the efficacy of the FOCUS ADHD in treatment adherence, symptom control and psychoeducation for the follow-up of ADHD patients. This implementation aims to involve health professionals and ADHD patients into a participatory, dynamic social processes to evaluate the proposed solution. In addition to the implementation of FOCUS ADHD, this study will also evaluate the impact on granting a discount on the purchase of psychostimulant medication. In Brazil, with some state exceptions, access to psychostimulant medication for ADHD treatment is not offered free of charge to the population by the State. Therefore, \the patient needs to pay out-of-pocket cost to acquire ADHD medications. The cost and access to medication is a significant factor for treatment abandonment. Thus, we intend to evaluate whether the granting of a significant discount on the acquisition of medication can have a positive impact on the treatment of adult patients with ADHD. This is three arms randomized clinical trial involving 60 adult ADHD patients that will be monitored for 3 months. One arm will be evaluating the impact of FOCUS ADHD app on treatment adherence. A second arm will be evaluating the FOCUS ADHD App plus the eligibility to receive the discount on the medication purchase. The third Arm will be based on current practices of ADHD patient follow up (treatment as usual). The patients will be recruited through public calls led by the Attention Deficit/Hyperactivity Program (PRODAH-A) of the Hospital de Clínicas de Porto Alegre (HCPA), Federal University of Rio Grande do Sul (UFRGS), Brazil. The primary outcomes will be evaluated by comparing the groups that used the mHealth FOCUS ADHD tool and the control that will not use them in the application. The primary outcome are:

* Adherence to pharmacological treatment of ADHD: Assess whether the use of the FOCUS ADHD application as a monitoring and education tool: (1) Increases by 10% the ADHD pharmacological treatment in adult patients compared to the control intervention. (2) Evaluate if a discount concession on ADHD pharmacological treatment increases by 20% the treatment adherence compared to the control intervention.
* ADHD knowledge and psychoeducation: Evaluate whether the use of the FOCUS ADHD application as a psychoeducation tool produces a at least 10% greater increase on knowledge about ADHD versus the control group.

Secondary outcomes will be evaluated exclusively with FOCUS ADHD application users. It will be evaluated levels of adoption, retention, and usability of the FOCUS ADHD application by enrolled participants. For the secondary outcomes evaluation, the following aspects will be analysed:

1. Adoption: Assess whether at least 50% patients have established with their respective physicians a collaborative network of ADHD monitoring through the FOCUS ADHD application. Assess whether at least 50% patients registered the medications in the Tasks and Medications icon. Assess whether at least 50% of patients filled out the ASRS symptom assessment at least once in the application. To verify whether at least 50% of patients-maintained access at least once a week to the news and psychoeducation contents of FOCUS in the period evaluated.
2. Retention: Examine whether at least 50% of patients who used the FOCUS ADHD app recorded at least 80% of days taking the daily medication on the evaluation period.
3. Usability assessment by implementing the User Version of the Mobile Application Rating Scale (uMARS). Obtain an average minimum score greater than or equal to 3 in the evaluations performed by users.

ELIGIBILITY:
Inclusion Criteria:

* Subject is willing and able to comply with all requirements of the study;
* Subject is able to provide written consent;
* Subject has a diagnosis of ADHD according to DSM-5;
* age 45 < 18 years;
* own smartphone;
* ASRS score at diagnosis ≥ 24
* Subject accepts usage of pharmacological treatment for ADHD during the study;

Exclusion Criteria:

* patients with any unstable or chronic clinical disease without adequate treatment, notified arterial hypertension, heart, kidney or liver diseases;
* presence of unstable psychiatric comorbidities requiring immediate treatment such as depression at risk of suicide or substance abuse/dependence, including anxiety and bipolar disorder. current or past history of psychosis;
* Patients with incomplete high school

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 73 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Adherence to pharmacological treatment of ADHD | Treatment adherence will be monitored through weekly telephone contact. Week 1 to 12.
  Treatment adherence will be calculated using the medication possession ratio (MPR) as the total number of days provided for the medication, divided by the number of days between the first and last dispensation; An 80% MPR will be used as the cut-off point between adherence and non-adherence. For the group that includes the discount on medication it will be evaluated the frequency of registration in the medication intake in the FOCUS ADHD application database as eligibility criteria for the discount concession.
ADHD Knowledge Change | The participants knowledge on ADHD should be carried out in two moments to evaluate the change or not of participants ADHD knowledge. At the beginning of the study on the baseline assessment and at the end of the follow-up period (Week 12)
  This is a questionnaire created in order to identify participants awareness about ADHD and the degree of information/misinformation about the disease and its management.

SECONDARY OUTCOMES:
FOCUS ADHD Adoption | End of the follow up period (Week 12)
  It will be analysed on app database if participants allocated to the app intervention arms, downloaded the app and established with their respective physician a collaborative network of ADHD monitoring through the FOCUS ADHD application, registered the medications in the Tasks Medications icon, filled out the ASRS symptom assessment in the application and accessed at least once a week the psychoeducation contents on the evaluated period.
FOCUS ADHD Retention | Weekly assessments Week 1 to Week 12
  It will be evaluated in the FOCUS ADHD database if participants recorded their treatment plan on the app and checked their medication intake in the tool.
FOCUS ADHD Usability | End of the follow up period (Week 12)
  Usability will be evaluated by implementation of the User Version of the Mobile Application Rating Scale (uMARS). This questionnaire will sent for participants using the FOCUS ADHD App. uMARS evaluates the Usability of digital solutions according to the following dimensions: engagement, functionality, aesthetics, information and subjective quality. It has 20 items divided scales of 5 points. Subscales are calculated by the average of the respective domain items. A total uMARS score is calculated by the average of all subdomains, while subjective quality is calculated by the average of its related subitems.

CONTACTS AND LOCATIONS:
Overall Officials: Luis Augusto P Rohde, MD-PhD, Principal Investigator — Hospital das Clínicas de Porto Alegre
Locations (1):
- Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Carvalho LR, Haas LM, Zeni G, Victor MM, Techele SP, Marrone Castanho J, Meneghetti Coimbra I, de Freitas de Sousa A, Ceretta N, Garrudo A, Grevet EH, Rohde LA. Evaluation of the effectiveness of the FOCUS ADHD App in monitoring adults with attention-deficit/hyperactivity disorder. Eur Psychiatry. 2023 Jun 21;66(1):e53. doi: 10.1192/j.eurpsy.2023.2422. PMID 37341028
- See also: Published Article at European Psychiatry — https://www.cambridge.org/core/journals/european-psychiatry/article/evaluation-of-the-effectiveness-of-the-focus-adhd-app-in-monitoring-adults-with-attentiondeficithyperactivity-disorder/D472E6CACE7D5AFB00CA40DDE898A6A7

DOCUMENTS (2):
  • Study Protocol (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT05551689/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-25): https://cdn.clinicaltrials.gov/large-docs/89/NCT05551689/SAP_001.pdf